CLINICAL TRIAL: NCT04769804
Title: Detection of IL1-7A and IL-17F Gene Polymorphism in Pityriasis Versicolor and Its Relation to Susceptibility to Infections.
Brief Title: Gene Polymorphism in Tinea Versicolor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer of dermatology, Kasr El Aini Hospital
Other Study IDs: PolymorphismTV
Record Dates: First submitted 2021-02-21; First posted 2021-02-25 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Pityriasis Versicolor
MeSH Terms: conditions — Tinea Versicolor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with recurrent pityriasis versicolor
- Healthy age and sex-matched controls

SUMMARY:
Blood samples will be taken from cases presenting with recurrent tinea versicolor , after confirmation of diagnosis by wood's light and KOH examination, for the detection of gene polymorphism in IL17 A and IL17 F.

In addition , serum samples from patients and controls will be tested for 25(OH)2 D3

ELIGIBILITY:
Inclusion Criteria:

* - Patients with recurrent pityriasis versicolor (active now) and not taking treatment for it.
* Patients of both genders.
* Age ≥18 years old.

Exclusion Criteria:

* - Patients with other cutaneous diseases.
* Patient's having dandruff (scaly scalp) even if not symptomatizing.
* Pregnant and lactating females, children, prisoners, cognitively impaired or mentally disabled subjects.
* Patients with autoimmune diseases.
* Patients with immunodeficiency diseases.
* Immunosuppressed patients e.g. HIV, diabetics, organ transplant, malignancy, patients taking immunosuppressive drugs e.g. chemotherapy, cortisone.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with history of disseminated TV, with 2 or more episodes of TV per year.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
IL 17A gene polymorphism | 6months-1 year
  IL 17A
IL 17 F gene polymorphism | 6months-1 year
  IL 17 F

SECONDARY OUTCOMES:
Vitamin D | 6months-1 year
  Serum 25(OH)2 D3

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Hospital, Cairo university, Cairo, El Manial, Egypt